CLINICAL TRIAL: NCT04879277
Title: Etude de l'INflammation systémique de Bas GRade Chez Les Patients Adultes Atteints de PHénylcétonurie
Brief Title: Study of Low-grade Systemic Inflammation in Adult Patients With Phenylketonuria
Acronym: INGRAPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DR210098; 2021-A01035-36 (Other: IdRCB)
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Phenylketonuria
Keywords: Low grade inflammation; Cardiovascular; Phenylketonuria
MeSH Terms: conditions — Phenylketonurias | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: One group of healthy subject and one group of patient with phenylketonuria. Primary objective is to compare inflammation profile between the two groups through cytokine assay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subject (Other): The intervention, specific to the study, is to take blood samples on patients healthy volunteers.
  Healthy subject will be paired to patient with phenylketonuria according to body mass index and sex.
  Interventions: Biological: Blood samples
- Patient with phenylketonuria (Other): The intervention, specific to the study, is to take blood samples on patients with phenylketonuria
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — Plasmatic cytokine and plasmatic CRP assay will be realised using luminex in both arms. IL2, IL10,INF gamma, IL, IL6, ILB, TNF alpha will be analysed.
  Other Names: Plasmatic Cytokine and plasmatic CRP assay

SUMMARY:
Patient suffering from phenylketonuria have chronic hyperphenylalaninemia. Hyperphenylalaninemia is known to be toxic to central nervous system and cardiovascular system in particular through oxydative stress.

In this context, research of low grade systemic inflammation through cytokine assay appears legitimate.

The primary outcome of this study is to describe inflammation profile of patients with phenylketonuria.

DETAILED DESCRIPTION:
Phenylketonuria (PKU) is a metabolic hereditary disease due to lack of activity of phenylalanine hydroxylase. This lack of activity whom origin is genetic, results in chronic hyperphenylalaninemia, toxic to central nervous system and cardiovascular system. Without treatment, PKU is responsible for mental retardation in children.

PKU is subject to systematic screening at birth and if diagnosis is confirmed a specific diet controlled in phenylalanine is prescribed for infant. This diet allows a neurodevelopment as closed as healthy infant. Despite this diet, neurological and systemic complications are more often reported at adult age. It is therefore recommended to follow patient regularly in order to search for those complications.

In a PKU murine model, it has been shown (cf references) that a low grade systematic inflammation exists and was reversible after dietetic treatment using glycomacropeptide (through a probiotic effect of this protein naturally phenylalanine free). Existence of this low grade systematic inflammation, evaluated by plasmatic cytokine screening (TNF alpha IL2, IL6, IL10, IFNgamma, IL1Alpha, IL1Beta and protein C reactive) has not been proven in humans to date.

Primary outcome of this study is to characterize this low grade systemic inflammation profile in patient with PKU.

ELIGIBILITY:
Inclusion Criteria (patient with PKU)

* Age >/= 18 years old
* Phenylketonuria diagnosis
* Fasting condition
* Registered with a social security system
* Patient consent

Inclusion Criteria (healthy volunteer)

* Age >/= 18 years old
* No metabolic condition
* Fasting condition
* Paired to patient with phenylketonuria already included according to age, sex and BMI class
* Registered with a social security system
* Volunteer consent

Exclusion Criteria, common to healthy volunteer and patient with phenylketonuria

* Pregnant and lactating women
* Subject to legal protection measures.
* Chronic or acute inflammatory disease
* Fever on inclusion
* Undergoing anti inflammatory treatment
* Surgery in the previous months
* Diabetes
* Included in other therapeutic trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of pro-inflammatory cytokines | At the inclusion
  Plasmatic pro-inflammatory cytokine assay in PKU patients and healthy subjects.
Plasma concentrations of CRP | At the inclusion
  Plasmatic CRP assay in PKU patients and healthy subjects.

SECONDARY OUTCOMES:
Plasma concentrations of phenylalanine | At the inclusion
  Plasmatic phenylalanine assay in PKU patients
Plasma concentrations of tyrosine | At the inclusion
  Plasma tyrosine assay in PKU patients

CONTACTS AND LOCATIONS:
Overall Officials: François MAILLOT, MD-PhD, Study Director — University Hospital, Tours
Locations (2):
- France (2):
  - Clinical investigation center, University Hospital, Tours, Tours
  - Internal Medicine Service, University Hospital, Tours, Tours

REFERENCES:
- [Background] Solverson P, Murali SG, Brinkman AS, Nelson DW, Clayton MK, Yen CL, Ney DM. Glycomacropeptide, a low-phenylalanine protein isolated from cheese whey, supports growth and attenuates metabolic stress in the murine model of phenylketonuria. Am J Physiol Endocrinol Metab. 2012 Apr 1;302(7):E885-95. doi: 10.1152/ajpendo.00647.2011. Epub 2012 Jan 31. PMID 22297302
- [Background] van Spronsen FJ, van Wegberg AM, Ahring K, Belanger-Quintana A, Blau N, Bosch AM, Burlina A, Campistol J, Feillet F, Gizewska M, Huijbregts SC, Kearney S, Leuzzi V, Maillot F, Muntau AC, Trefz FK, van Rijn M, Walter JH, MacDonald A. Key European guidelines for the diagnosis and management of patients with phenylketonuria. Lancet Diabetes Endocrinol. 2017 Sep;5(9):743-756. doi: 10.1016/S2213-8587(16)30320-5. Epub 2017 Jan 10. PMID 28082082
- [Background] Boulet L, Besson G, Van Noolen L, Faure P; ECOPHEN Study Group; Maillot F, Corne C. Tryptophan metabolism in phenylketonuria: A French adult cohort study. J Inherit Metab Dis. 2020 Sep;43(5):944-951. doi: 10.1002/jimd.12250. Epub 2020 Jun 4. PMID 32392388
- [Background] Stroup BM, Nair N, Murali SG, Broniowska K, Rohr F, Levy HL, Ney DM. Metabolomic Markers of Essential Fatty Acids, Carnitine, and Cholesterol Metabolism in Adults and Adolescents with Phenylketonuria. J Nutr. 2018 Feb 1;148(2):194-201. doi: 10.1093/jn/nxx039. PMID 29490096
- [Background] Matalon R, Surendran S, McDonald JD, Okorodudu AO, Tyring SK, Michals-Matalon K, Harris P. Abnormal expression of genes associated with development and inflammation in the heart of mouse maternal phenylketonuria offspring. Int J Immunopathol Pharmacol. 2005 Jul-Sep;18(3):557-65. doi: 10.1177/039463200501800316. PMID 16164837
- [Result] Giret C, Dos Santos Y, Blasco H, Paget C, Gonzalez L, Tressel N, Dieu M, Bigot A, Gissot V, Audemard-Verger A, Maillot F. No evidence for systemic low-grade inflammation in adult patients with early-treated phenylketonuria: The INGRAPH study. JIMD Rep. 2023 Oct 4;64(6):446-452. doi: 10.1002/jmd2.12366. eCollection 2023 Nov. PMID 37927482